CLINICAL TRIAL: NCT04020198
Title: A Pilot Biomarker Study Assessing Alpha-synuclein Aggregates Across Biofluid Reservoirs in Patients With Synucleinopathies
Status: Terminated | Type: Observational
Why Stopped: The assay under investigation did not show evidence of accurately detecting alpha-synuclein in specimens collected in the study other than CSF and the intention of the study was to identify less invasive ways to measure alpha-synuclein.
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Carine Maurer, Assistant Professor, Stony Brook University
Other Study IDs: SNCA 1355881
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Rapid Eye Movement Sleep Behavior Disorder; Normal Pressure Hydrocephalus
Keywords: Alpha-synuclein
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; REM Sleep Behavior Disorder; Hydrocephalus, Normal Pressure; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — CSF, plasma, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Parkinson's Disease: Subjects who have a PD diagnosis
  Interventions: Other: Biomarker assay
- Multiple System Atrophy: Subjects who have an MSA diagnosis
  Interventions: Other: Biomarker assay
- Age-matched controls: Subjects who do not have a diagnosed parkinsonian disorder
  Interventions: Other: Biomarker assay
- Rapid Eye Movement Sleep Behavior Disorder (RBD): Subjects who have a diagnosis of RBD
  Interventions: Other: Biomarker assay
- Normal Pressure Hydrocephalus: Subjects who are prescribed a lumbar puncture to treat normal pressure hydrocephalus
  Interventions: Other: Biomarker assay

INTERVENTIONS:
Other: Biomarker assay — Biomarker assay will be used to quantify levels of misfolded alpha-synuclein aggregates in biofluid samples from patients with Parkinson's disease, multiple system atrophy, rapid eye movement sleep behavior disorder, normal pressure hydrocephalus and controls.

SUMMARY:
This will be an observational study looking at clinical and biomarker characteristics in patients with Parkinson's Disease (PD), Multiple System Atrophy (MSA), Rapid Eye Movement Sleep Behavior Disorder (RBD), Normal Pressure Hydrocephalus and matched controls. Saliva, plasma, serum, urine, and cerebrospinal fluid (CSF) samples will be collected from participants.

DETAILED DESCRIPTION:
This is an observational study looking at clinical and biomarker characteristics in patients with Parkinson's disease (PD), Multiple System Atrophy (MSA), Rapid Eye Movement Sleep Behavior Disorder (RBD), Normal Pressure Hydrocephalus (NPH) and matched controls. Saliva, plasma, serum, urine, and cerebrospinal fluid samples will be collected from participants. Samples will be assessed for levels of misfolded alpha-synuclein aggregates. Clinical characteristics will also be assessed.

Misfolded alpha-synuclein aggregates have the potential to serve as an early biomarker for PD and MSA, increasing the ability to diagnose and treat individuals with these diseases earlier. This study examines the effectiveness of using a novel technique for distinguishing between different parkinsonian disorders by measuring small misfolded α-synuclein aggregates in different biofluids.

ELIGIBILITY:
For PD subjects:

Inclusion Criteria:

1. Age 50-75
2. Diagnosis of idiopathic PD as confirmed by a movement disorder specialist
3. Age of onset of motor symptoms between 50 - 75
4. Well-established response to dopaminergic agents and/or amantadine
5. Ability to complete questionnaires
6. Ability to provide informed consent
7. Willingness to go off parkinsonian medication for 12 hours prior to "off" assessment
8. Medical record includes a brain MRI taken within the past 12 months showing no evidence of a tumor or abscess

Exclusion Criteria:

1. Symptomatic (secondary) parkinsonism (ie. drug induced)
2. Atypical parkinsonian variants
3. History of cancer (except basal or squamous cell skin cancer) within 5 years
4. Known liver disease
5. Hematological disorders
6. History of stereotactic or ablative brain surgery
7. Treatment with an investigational drug or device within the last 30 days
8. Pregnancy
9. Inability to comply with or tolerate study procedures
10. Conditions precluding the safe performance of lumbar puncture (LP): use of anticoagulants and hematologic abnormalities (INR>1.3;platelet count <80,000)

MSA Subjects:

Inclusion Criteria:

1. Age 50-75
2. Age of onset of motor symptoms between 50-75
3. Diagnosis of probable or possible MSA as confirmed by a movement disorders specialist
4. Ability to complete questionnaires
5. Ability to provide informed consent
6. Willingness to go off parkinsonian medications for 12 hours prior to "off" assessment
7. Medical record indicates a brain MRI taken within the past 12 months showing no evidence of a tumor or abscess

Exclusion Criteria

1. Symptomatic (secondary) parkinsonism (ie. drug induced)
2. History of cancer (except basal or squamous cell skin cancer) within 5 years
3. Known liver disease
4. Hematological disorders
5. History of stereotactic or ablative brain surgery
6. Treatment with an investigational drug or device within the last 30 days
7. Pregnancy
8. Inability to comply with or tolerate study procedures
9. Conditions precluding the safe performance of lumbar puncture (LP): use of anticoagulants and hematologic abnormalities (INR>1.3;platelet count <80,000)

For RBD Subjects:

Inclusion Criteria:

1. Age 50-75
2. Diagnosis of RBD using current consensus criteria
3. Ability to provide informed consent
4. Ability to complete questionnaires
5. Medical record indicates a brain MRI taken within the past 12 months showing no evidence of a tumor or abscess

Exclusion Criteria

1. Signs for symptoms suggestive of parkinsonian disorder
2. History of cancer (except basal or squamous cell skin cancer) within 5 years
3. Known liver disease
4. Hematological disorders
5. History of stereotactic or ablative brain surgery
6. Treatment with an investigational drug or device within the last 30 days
7. Pregnancy
8. Inability to comply with or tolerate study procedures
9. Conditions precluding the safe performance of lumbar puncture (LP): use of anticoagulants and hematologic abnormalities (INR>1.3;platelet count <80,000)

For NPH:

Inclusion Criteria:

1. Age 50-75
2. Scheduled to undergo an LP to evaluate diagnosis of NPH at Stony Brook Neurological Associates
3. Ability to complete questionnaires
4. Ability to provide informed consent

Exclusion Criteria:

1. History of cancer (except basal or squamous cell skin cancer) within 5 years
2. Known liver disease
3. Hematological disorders
4. History of stereotactic or ablative brain surgery
5. Treatment with an investigational drug or device within the last 30 days
6. Pregnancy
7. Inability to comply with or tolerate study procedures
8. Conditions precluding the safe performance of lumbar puncture (LP): use of anticoagulants and hematologic abnormalities (INR>1.3;platelet count <80,000)

For Controls:

Inclusion Criteria:

1. Age 50-75
2. Scheduled to undergo an LP at Stony Brook Neurological Associates
3. Ability to complete questionnaires
4. Ability to provide informed consent

Exclusion Criteria:

1. Signs or symptoms suggestive of parkinsonian disorder
2. History of rapid eye movement (REM) Sleep Behavior Disorder (RBD)
3. History of cancer (except basal or squamous cell skin cancer) within 5 years
4. Known liver disease
5. Hematological disorders
6. History of stereotactic or ablative brain surgery
7. Treatment with an investigational drug or device within the last 30 days
8. Pregnancy
9. Inability to comply with or tolerate study procedures
10. Conditions precluding the safe performance of lumbar puncture (LP): use of anticoagulants and hematologic abnormalities (INR>1.3;platelet count <80,000)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with PD, MSA, RBD, NPH and controls
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Compare levels of misfolded alpha-synuclein aggregates in participants with PD, MSA, RBD, NPH and controls | 3 weeks
  Levels of misfolded alpha-synuclein in CSF, serum, plasma, saliva, and urine will be quantified using the protein misfolding cyclic amplification (PMCA) technology

SECONDARY OUTCOMES:
Investigate the relationship between levels of misfolded alpha-synuclein aggregates and disease severity in PD and MSA | 3 weeks
  Levels of misfolded alpha-synuclein aggregates will be quantified using the PMCA technology. PD and MSA disease severity will be assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the Unified Multiple System Atrophy Rating Scale (UMSARS), respectively. All groups will receive the MDS-UPDRS III and the RBD Questionnaire.
Investigate the relationship between levels of misfolded alpha-synuclein aggregates across different biofluid reservoirs, including CSF, serum, plasma, saliva, and urine | 3 weeks
  Levels of misfolded alpha-synuclein in the different biofluid reservoirs will be quantified using the PMCA technology

CONTACTS AND LOCATIONS:
Overall Officials: Carine W. Maurer, MD, PhD, Principal Investigator — Stony Brook University Medical Center
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Identifiers will be removed from participant data or biospecimens. After such removal, the information or biospecimens may be used for future research studies.